CLINICAL TRIAL: NCT02796612
Title: Empathy and Standard Diagnostic Procedures in an Outpatient Breast Clinic Might Not be Enough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EK261/12
Record Dates: First submitted 2015-07-17; First posted 2016-06-13 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Anxiety
Keywords: anxiety; breast cancer, suspected; breast biopsy; empathy; standardized and structured information; anxiety reduction
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (Active Comparator): Patients receive the current standard of care and are asked to answer the questionnaires mentioned below.
  Interventions: Other: no intervention
- Intervention group (Experimental): Patients receive the current standard of care and are asked to answer the questionnaires mentioned below.
  Additionally, delivery of a take-home brochure to the patients during the first visit is planned. The biopsy is explained to the patient and performed by a psychological trained physician. Patient care by a psychologically trained physician is performed in the sense that patients are informed about their biopsy result by a specifically trained physician.
  Interventions: Other: no intervention; Behavioral: delivery of a take-home brochure; Behavioral: patient care by a psychologically trained physician

INTERVENTIONS:
Other: no intervention — Patients do not receive any interventions but are treated according to current standard of care.
Behavioral: delivery of a take-home brochure — Content of brochure is dealing with symptoms, as well as mammographic and ultrasound findings, which need further investigation, will be addressed. The procedure of the breast biopsy itself will be explained in detail. The time in which the histological diagnosis can be expected will be indicated and follow up in case of a benign histology and the necessary therapy in case of breast cancer will be addressed.
  Arms: Intervention group
Behavioral: patient care by a psychologically trained physician — The physicians who perform the biopsies will be instructed by means of a psychological training how to give structured and standardized information in order not only to inform comprehensively, but also to meet the patients' emotional needs.
  Arms: Intervention group

SUMMARY:
The project investigates prospectively whether anxiety in the context of breast biopsy can be reduced by the planed intervention (take-home brochure and structured and standardized information given by a psychologically trained physician who performs the biopsy).

DETAILED DESCRIPTION:
The fact having to have a breast biopsy taken due to suspected breast cancer is an emotionally exceptional situation not only because of the threat to be diagnosed of cancer but also because the breast is perceived as a symbol of womanhood, sexuality and motherhood.

Time, however, is scarce in a busy outpatient setting. Nevertheless doctors and nurses at the outpatient breast clinic University Hospital Basel are empathetic and try to address anxiety and give emotional support before, during, and after a necessary breast biopsy. Study findings, however suggest, that the level of anxiety, pain and discomfort associated with breast biopsies is considerable, which might not be sufficiently controlled by empathy alone but might be reduced by giving structured and standardized information.

The investigators hypothesize that the planned intervention reduces the level of anxiety in patients going for breast biopsy and thus is superior to the current standard of diagnostic procedures.

The project focuses on improving the patients' knowledge about the procedure of breast biopsy and on meeting their emotional needs to reduce anxiety related to the biopsy by giving structured and standardized information. Additionally the project investigates whether patients diagnosed with breast cancer have a higher level of anxiety than patients with benign breast disease. Furthermore the study assesses how precisely the physicians, who perform the biopsy, appraise the patients' perception of anxiety, pain and satisfaction related to the breast biopsy.

The primary objective is to demonstrate that the intervention reduces the patients' anxiety compared to the standard of care.

The intervention consists of (1) handing out a take-home brochure to the patient as well as (2) providing structured standardized information about the biopsy by the physician who performs the biopsy and who underwent psychological training for this purpose.

Secondary objectives are:

Does the intervention reduce anxiety during and after biopsy? Is there a correlation of the level of anxiety and the histological diagnosis of breast cancer? Does the waiting time between the procedure and the histological diagnosis have any influence on the level of anxiety? How is the patient's perception of pain during and after the biopsy? Is there a correlation between the patient's perception of pain and anxiety and the physicians' impression of the patient's perception? Is the patient satisfied with the additional take-home brochure and / or the structured and standardized information giving? This is a prospective study to evaluate anxiety before and after the implementation of a structured intervention to reduce anxiety related to breast biopsy.

Eligible are women who speak and understand German and will need a skin biopsy, core biopsy or a vacuum assisted biopsy.

Women receiving a fine needle aspiration, examination of a pathologic nipple secretion, and abscess evacuation will be excluded.

Women who do not understand or do not speak the German language will be excluded.

Demographics and relevant baseline variables will be summarized for both groups of patients. Categorical data will be presented as frequencies and percentages. For continuous variables, the lower and upper quartile as well as the median will be presented. Baseline characteristics of the two groups will be compared using the proportion test for categorical variables and the Welch two-sample t-test for continuous variables.

Anxiety of patients will be measured at four points in time with State-Trait Anxiety Inventory (STAI): before and after biopsy as well as before and after the communication of the diagnosis. The difference in STAI score between patients receiving standard of care and patients with intervention will be compared using Wilcoxon's rank sum test (Mann-Whitney test) at a significance level of α = 0.05. The results of the questionnaires will be reported as estimates together with the 95% confidence interval. Secondary objectives will be assessed using non-parametric tests if appropriate.

Sample size was estimated to be able to detect a significant difference in anxiety measured by the State-Trait Anxiety Inventory (STAI) score (Spielberger, Consulting Psychologists Press (CPP) 1983) between the group receiving standard of care and the intervention group. In a recent study, Flory et al. (Flory and Lang) reported a mean STAI score of 48 points for breast biopsy patients which were used here to simulate data for the control group. By assuming an effect size of 5 score points, a mean score of 43 points was used for the patients with intervention. The scores of both groups were assumed to be normally distributed with a standard deviation of 11.9.

Sample size was calculated with a semi-parametric resampling method. Each sample size ni, was evaluated by simulating R=999 times ni individual patients from the above distributions. The scores of the two groups were compared using Wilcoxon's signed-rank test at a significance level of α = 0.05. Sample size was set to ensure at least a power, 1 - β, of 0.9.

For this study, totally 334 patients should be recruited to ensure 250 evaluable patients considering a drop-out rate of 25 %.

ELIGIBILITY:
Inclusion Criteria:

* women who speak and understand German
* women who will need a skin biopsy, core biopsy or a vacuum assisted biopsy.

Exclusion Criteria:

* women receiving a fine needle Aspiration
* women receiving an examination of a pathologic nipple secretion
* women receiving an abscess evacuation
* women who do not speak and understand German

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Reduction of level of anxiety compared between arm 'no intervention' and arm 'intervention' as measured via questionnaires | up to 19 months

SECONDARY OUTCOMES:
level of anxiety in the intervention group during and after biopsy measured via questionnaires | up to 19 months
correlation of the level of anxiety and the histological diagnosis of breast cancer measured via questionnaires | up to 19 months
perception of pain during and after biopsy measured via pain score | up to 19 months
influence of waiting time between biopsy and histological diagnosis on the level of anxiety measured via questionnaires | up to 19 months
correlation of patient's perception of pain and anxiety and physician's impression of patient's perception measured by questionnaires | up to 19 months
patient's satisfaction with additional information concerning biopsy measured by Visual Analog Scale | up to 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Zanetti, PD Dr. MD, Principal Investigator — Claraspital Basel
Locations (3):
- Switzerland (3):
  - University Hospital of Basel, Basel, Canton of Basel-City
  - Claraspital, Basel, Canton of Basel-City
  - GZO Wetzikon, Wetzikon, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Machacek M, Urech C, Tschudin S, Werlen L, Schoenenberger CA, Zanetti-Dallenbach R. Impact of a brochure and empathetic physician communication on patients' perception of breast biopsies. Arch Gynecol Obstet. 2023 Nov;308(5):1611-1620. doi: 10.1007/s00404-023-07058-w. Epub 2023 May 20. PMID 37209201